CLINICAL TRIAL: NCT03919903
Title: Parent's Knowledge, Attitude and Practices Towards Oral Health of Their Children With Primary Dentition: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Ahmed Mohamed Helal, General Dentist, Cairo University
Other Study IDs: Parent's Oral Health Knowledge
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Oral Health Knowledge

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study aims to assess Parents Knowledge, Attitude and Practices towards Oral Health of their Children with Primary Teeth.

DETAILED DESCRIPTION:
Dental caries is a chronic slowly progressing localized destruction of dental hard tissues by the acidic products formed as result of carbohydrates fermentation by bacteria due to disturbance in equilibrium between tooth minerals and plaque products through time. (Trindade et al., 2014) It's a worldwide disease affecting all ages both sexes with different socioeconomic levels. Dental caries commonly affects children and adversely affects their quality of life and so their weight and growth if left untreated (Gokhale and Nuvvula, 2015). The environmental factor is a very valuable factor affecting dental caries especially the mother and the family as whole, the family habits are directly influencing their children (Suma G and Anisha P, 2017). As parents are the primary decision makers for children and their first role models, their oral health knowledge, attitude and practice as well as habits influence their children (Dikshit et al., 2018).

There is lack of data about parent's oral health knowledge, attitude and practice and their implications on their children in Egypt.

Acquiring information about oral health knowledge of parents, will help identifying those children who are at risk of dental caries consequently it will be possible to offer the proper preventive and curative measures for them.

So, we need to know the effect of oral health knowledge, attitude and practice (KAP) of parents on caries prevalence of their children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and their parents.
* Children with primary dentition.

Exclusion Criteria:

* Parents refuse to participate.

Ages: 1 Year to 8 Years | Sex: All
Age Groups: Child
Study Population: Parents of children with primary dentition
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Parents Oral Health Knowledge, Attitude and Practice (KAP) | one year
  Questionnaire is the measurement tool for the primary outcome, questionnaires will be admitted to the parents in the waiting area of the diagnostic clinic of Pediatric dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.The questionnaire consists of 28 questions; 10 related to knowledge, 6 to attitude, 8 to practice and 4 general questions. The response will be assessed by using a scoring system, where scores are based on correct answers. For the knowledge and practice items, the right answer is coded as 1 and the wrong answer as 0. For attitude items score 1 indicates a positive attitude, while score 0 indicates a negative attitude. The individual scores will then be summed up to yield a total score. Maximum possible score will be 10, 6 and 8 for KAP respectively. Mean Score of <40% and≥ 40 % are considered as inadequate and adequate performance respectively. (Dikshit et al., 2018) The questionnaire was translated in Arabic language.

SECONDARY OUTCOMES:
Caries Prevalence in their children | one year
  Caries Prevalence in the children will be assessed by clinical examination. Examination will be performed at the diagnostic clinic of the Pediatric dentistry department, Faculty of Dentistry, Cairo University. Patient assessment chart will be used for recording the oral assessment data. The oral assessment of every child will be done by a single operator under good lighting condition using mouth mirror and probe to detect the presence of carious (whether smooth or pits and fissure caries), missed (extracted) and filled teeth (Cypriano et al., 2005).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pediatric Dentistry and Dental public Health, Cairo University, Cairo, Egypt

REFERENCES:
- See also: Evaluation of Knowledge, Attitude and Practices of Parents toward their Children Oral Health Compared with their Dental Caries status — https://www.nepjol.info/index.php/bjhs/article/view/20943
- See also: Knowledge, Attitudes And Practices of Parents Regarding Oral Health and Its Correlation with Dental Caries Status of Their Children: A Cross Sectional Study — https://www.researchgate.net/publication/304764240_Knowledge_Attitudes_And_Practices_of_Parents_Regarding_Oral_Health_and_Its_Correlation_with_Dental_Caries_Status_of_Their_Children_A_Cross_Sectional_Study